CLINICAL TRIAL: NCT05853705
Title: Strong Hearts: A Remote, App-Enabled, Exercise Program for Patients With Congenital Heart Disease
Brief Title: Strong Hearts: A Remote, App-Enabled, Exercise Program for Patients With Congenital Heart Disease (Strong Hearts App)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low participation rate
Sponsor: Duke University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00111958
Record Dates: First submitted 2023-04-14; First posted 2023-05-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Congenital Heart Disease
Keywords: Child; Adult
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise Group (Experimental): Participants will participate in a remote, app-enabled exercise program consisting of strength and aerobic exercises for four to twelve weeks. They will perform the exercises 3-5 times a week at home guided by exercise videos in the app. The exercise sessions will increase in frequency throughout the training regimen. The videos will include athletes demonstrating how to perform each exercise safely, and provide tips for optimal form and breathing. Participants will wear wearable fitness trackers and monitor their heart rates during exercise sessions.
  Interventions: Behavioral: Strong Hearts Exercise Program

INTERVENTIONS:
Behavioral: Strong Hearts Exercise Program — The participant will either begin at the easiest variation of each strength exercise (level A), or will be placed at a specific level for each strength exercise based on their assessment with physical therapy. Participants can progress to the next level of difficulty of a specific strength exercise based on their rating of perceived exertion (RPE) with the opportunity to move to the next level if they have RPE score of 6 or less and if their heart rates are at goal. Each participant will be provided with heart rate ranges based on the heart rate reserve (HRR) method using their baseline resting and peak heart rates obtained during their cardiopulmonary exercise testing (CPET) or percent predicted heart rate based on age if CPET is not available. HRR goals will be set individually for patients and adjusted per protocol to guide effort.

SUMMARY:
The overall goal of this program is to create a remote, mobile application enabled exercise program for patients with Congenital Heart Disease (CHD). Pilot trials will consist of a remote exercise program with app-embedded exercise modules designed to promote and encourage safe and healthy exercise habits across a range of CHD anatomies. This app-enabled program will allow for real time data collection integrating wearable devices, as well as compliance and safety monitoring to enhance research capabilities. The app-enabled program will be versatile and may be applied in the future to patients with non-cardiac conditions.

ELIGIBILITY:
Inclusion Criteria:

* Repaired or unrepaired Congenital Heart Disease (CHD)
* Between ages 10 and 50, inclusive, at time of consent
* Android or Apple smartphone that meets the operating systems below with the ability to download applications from either Google Play or the Apple store

  * Android: 6.0 or higher
  * Apple: iPhone Operating System (iOS) 13 or higher

Exclusion Criteria:

* Physical or mental disabilities preventing exercise participation
* Uncontrolled systemic hypertension (symptomatic or greater than Stage 2 hypertension while on therapy)
* Poorly controlled arrhythmia
* Clinically unstable heart failure
* Known pregnancy at the time of enrollment

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Change in peak rate of oxygen volume consumption (VO2) on Cardiopulmonary Exercise Testing | Baseline, up to 12 weeks

SECONDARY OUTCOMES:
Change in Pediatric Cardiac Quality of Life Inventory | 1 year
  The Pediatric Cardiac Quality of Life Inventory generates 3 scores (total, disease impact subscale, and psychosocial impact subscale). Each subscale has a maximum of 50 points and their sums yields the total score. Higher scores indicate better perceived health-related quality of life.
Change in Short Form 36 (SF-36) Health Survey | 1 year
  The Short Form 36 Health Survey consists of 8 subscales (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health). The survey will be scored using the two step RAND scoring process. The first step scores each question on a scale from 0 (worst) to 100 (best) and represents the percentage of total possible score achieved. The second scoring step, takes the average of all the questions in each subscale to create the 8 scores.
Change in sit-to-stand test | Baseline, up to 12 weeks
Change in secondary Cardiopulmonary Exercise Testing outcome measures | Baseline, up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reid C Chamberlain, MD, MSCI, Principal Investigator — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No